CLINICAL TRIAL: NCT04669821
Title: A Multi-Center, Randomized, Open-Label, Propofol-Controlled Exploratory Clinical Study Evaluating Sedation of Intravenous Administration of HSK3486 Injectable Emulsion in ICU Patients Undergoing Long-Term Mechanical Ventilation
Brief Title: A Clinical Study Evaluating Sedation of Intravenous Administration of HSK3486 in ICU Patients Undergoing Long-Term Mechanical Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-206
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Sedation in Intensive Care
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental)
  Interventions: Drug: HSK3486
- Propofol (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — Loading Dose：0.1 mg/kg，Maintenance Dose：Maintenance is started at 0.3 mg/kg/h, and the dose can be adjusted up and down by 0.05-0.1 mg/kg/h.
  Arms: HSK3486
Drug: Propofol — Loading Dose：0.5 mg/kg，Maintenance Dose：Maintenance is started at1.5 mg/kg/h, and the dose can be adjusted up and down by 0.25-0.5mg/kg/h.
  Arms: Propofol

SUMMARY:
This is a multi-center, randomized, open-label, propofol-controlled exploratory clinical study. In this study, 20 ICU patients undergoing mechanical ventilation are expected to be enrolled and will be randomly assigned to the HSK3486 group and the propofol group in a 1:1 ratio. This study is not blinded as it is open-label.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require tracheal intubation for mechanical ventilation, with expected sedation duration of longer than 96 h;
2. Patients requiring a target RASS score of -1 to -2 for sedation;
3. Aged ≥ 18 and < 80 years old, with no gender requirement;
4. BMI ≥ 18 kg/m2 and ≤ 30 kg/m2;
5. The patients or their family members fully understand the objectives and significance of this study, and voluntarily participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Patients known to be allergic to eggs, soy products, opioids and their antidotes, and Propofol; patient having contraindications to Propofol, opioids and their antidotes;
2. Patients who have received propofol for more than 3 days in the ICU or in the general ward before being transferred to the ICU before signing informed consent form;
3. Patients having the following medical history or evidence of any of the following at screening, which may increase sedation/anesthesia risk:

   1. Cardiovascular system: New York Heart Association (NYHA) Class III and IV heart failure, Adams-stokes syndrome; acute coronary syndrome (ACS) that occurs within 6 months before screening; bradycardia requiring medication and/or heart rate ≤ 50 beats/min; a history of severe arrhythmia such as II-III degree atrioventricular block (excluding patients using pacemakers); acute and chronic myocarditis;
   2. Patients with hyperlipidemia: Defined as patients with TC ≥ 5.2 mmol/L or LDL-C ≥ 3.4 mmol/L at screening, or patients with severely increased blood pressure or blood glucose despite their blood lipid levels meeting the requirements, rendering the patients huge risk of cardiovascular diseases per the investigator's judgment; patients with acute pancreatitis;
   3. Patients with mental diseases (e.g., schizophrenia, depression) and cognitive dysfunction; grand mal epilepsy and convulsion; head injury, intracranial hypertension, cerebral aneurysm; Glasgow Coma Score (GCS) ≤ 12; SOFA Score > 9; past history of psychotropic and narcotic drug abuse; history of alcohol abuse within 3 months before screening; long-term use of psychotropic drugs;
   4. Patients with high paraplegia and general paralysis; patients with unstable hemodynamics;
   5. Severe hepatic and renal insufficiency (liver function: refer to child-pugh grade C; renal function: glomerular filtration rate eGFR ≤ 30 mL/(min•1.73 m2) [eGFR is calculated using the Modification of Diet in Renal Disease (MDRD) equation: eGFR = 175 × serum creatinine (SCr)-1.234 × age-0.179 × 0.79 (females)]; patients undergoing dialysis;
   6. Patients with an expected survival of less than 1 week;
   7. Other situations unsuitable for enrollment per the investigator's consideration.
4. Pregnant or breastfeeding females: women or men of child-bearing potential who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 1 month after the trial starts (including male subjects);
5. Have participated in any other clinical trials within 1 month prior to screening;
6. Other conditions that patients are judged by the investigator to be unsuitable for participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
Mean duration of qualified sedation | Within 96hours of administration
  the mean duration of RASS being in the range of -1 to -2 per hour during the study medication provided that no remedial medication is used

SECONDARY OUTCOMES:
Time to recovery | Within 24 hours after administration
  the time for the subject to recover from sedation to full recovery of consciousness (RASS ≥ 0) after discontinuation of drug administration.
Time to extubation | Within 24 hours after administration
  the time from intubation (applicable to patients who undergoes intubation after entering the ICU)/ICU admission (applicable to patients with intubation before entering the ICU) to extubation or the time from drug discontinuation to extubation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, China